CLINICAL TRIAL: NCT06950424
Title: Effect of Black Cumin Seed Oil on Cortisol, Stress and Quality of Life in Healthy Moderately-Stressed Adults
Brief Title: Effect of Black Cumin Seed Oil Supplementation on Cortisol, Stress and Mood
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shawn Talbott (Industry)
Responsible Party: Sponsor-Investigator, Shawn Talbott, PI, 3 Waves Wellness
Organization: 3 Waves Wellness (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: BlackSeedCortisol2025
Record Dates: First submitted 2025-04-21; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Stress; Mood
Keywords: stress; mood
MeSH Terms: interventions — Nigella sativa oil

STUDY DESIGN:
Intervention Model Description: Two arms - active supplement and placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement (Experimental): 500mg black cumin seed oil
  Interventions: Dietary Supplement: black cumin seed oil
- Placebo (Placebo Comparator): maltodextrin placebo
  Interventions: Dietary Supplement: black cumin seed oil

INTERVENTIONS:
Dietary Supplement: black cumin seed oil — 500mg of black cumin seed oil standardized for 3% thymoquinone)

SUMMARY:
The primary objective of this study will be to collect data to support the role of black cumin seed oil, also known as black seed oil (BSO), in moderating the stress response, including objective markers of stress (cortisol/DHEA) as well as subjective measures (mood/stress/sleep/beauty). The primary outcomes will be salivary cortisol, subjective stress, and psychological vigor.

Subjects will be recruited from among the clients of the Certified Mental Wellness Coaches (CMWCs) that have passed the digital badge course via Marietta College (https://www.credly.com/org/marietta-college/badge/certified-mental-wellness-coach-cmwc-online).

If volunteers meet the inclusion/exclusion criteria, they will review/sign the Informed Consent Form (ICF - attached) before any Baseline measurements are collected.

Because BSO is already known to deliver a wide range of potential health benefits, including anti-inflammatory, anti-oxidant, anti-diabetic, and immune-modulating effects - we expect to observe improvements on both subjective psychological and objective biochemical measures. Our primary outcome measures will be salivary cortisol and psychological mood state (POMS, including tension, mood, irritability, focus, fatigue, vigor and well-being).

DETAILED DESCRIPTION:
Black seed oil (BSO), derived from Nigella sativa, has been utilized in traditional medicine for centuries. Its active constituents, such as thymoquinone, nigellone, and other bioactive compounds, are associated with diverse pharmacological effects. Recent scientific investigations have confirmed its potential health benefits, particularly as a natural anti-inflammatory agent.

Historical records indicate the use of BSO as a spice and medicinal herb dating back at least 1,400 years. Traditional medicinal systems, including Unani, Islamic, and Ayurvedic medicine, recognize its wide-ranging therapeutic properties. Traditional uses of black seed oil include remedies for respiratory ailments, digestive disorders, and skin conditions. However, contemporary scientific investigations have provided more precise evidence of its effects on biochemical pathways involved in inflammation, cellular protection, energy metabolism, and stress responses.

Nigella sativa seeds are rich in various bioactive compounds, including:

* Thymoquinone (TQ): The most studied bioactive constituent with diverse pharmacological activities, including anti-inflammatory, antioxidant, antibacterial, and anticancer effects.
* Terpenes and Terpenoids: p-cymene, carvacrol, thymohydroquinone (THQ), dihydrothymoquinone (DHTQ), α-thujene, thymol, t-anethole, β-pinene, α-pinene, and γ-terpinene.
* Fatty Acids: Predominantly linoleic acid, oleic acid, and palmitic acid.
* Phytosterols: Notably, β-sitosterol and stigmasterol.
* Alkaloids: Including nigellicimine, nigellidine, and nigellamines.
* Polyphenols: Such as quercitrin and kaempferol.

Because of the diversity of bioactive compounds found in BSO, its historical usage as a "cure-all" across various traditional medicine systems, and our emerging understanding of its clinical utility against modern stress-related ailments, this study explores black seed oil's therapeutic potential and relevance to modern health challenges, particularly cortisol modulation and stress response.

We will be using a specific brand of black seed oil extract known as Thymoquin, which can be found in a large number of commercial dietary supplements = https://www.trinutra.com/thymoquin

Outcome Measures

Measurements will be made FOUR times: at Baseline and after study participants have consumed BSO or Placebo for 1 week, 4 weeks and 8 weeks:

Baseline, Week 1, and Week 4:

* Cortisol/DHEA Panel (4 measurements providing diurnal rhythm)
* Stress (10-item assessment of overall stress via Perceived Stress Scale; PSS)
* Mood (7 components of mood via Profile of Mood States; POMS)
* Sleep Quality (8 components of sleep via Pittsburgh Sleep Quality Index; PSQI)
* Beauty (5 components of beauty, skin health, and quality-of-life; BeautyQOL)
* Focus (2 components of attention via ADHD Self-Report Scale; ASRS)

Week 8:

* Stress (10-item assessment of overall stress via Perceived Stress Scale; PSS)
* Mood (7 components of mood via Profile of Mood States; POMS)
* Sleep Quality (8 components of sleep via Pittsburgh Sleep Quality Index; PSQI)

Methods

Salivary Cortisol/DHEA Cortisol is the major glucocorticoid produced in the adrenal cortex. Cortisol production has a circadian rhythm, with levels peaking in the early morning and dropping to lowest values at night. Levels rise independently of circadian rhythm in response to stress. In blood, only about 5-10% of cortisol is in its unbound or biologically active form. The remaining cortisol is bound to serum proteins. Unbound serum cortisol enters saliva via intracellular mechanisms; in saliva, the majority of cortisol remains unbound to protein. Studies consistently report high correlations between serum and salivary cortisol, indicating that salivary cortisol levels reliably estimate serum cortisol levels (https://www.sciencedirect.com/science/article/abs/pii/S0306453008002990; https://www.karger.com/Article/Abstract/118611)

During periods of stress, both cortisol and DHEA are secreted by the adrenal glands, but they often have opposing effects on the body. Cortisol is frequently referred to as the "stress hormone" because it helps mobilize energy reserves and regulate the body's response to stress, but excessive levels over time can contribute to inflammation and tissue breakdown. DHEA, on the other hand, acts as a counterbalance to cortisol: it can mitigate some of cortisol's negative impacts by supporting immune function and promoting tissue repair. The ratio of cortisol to DHEA is an important marker of physiological stress, and chronic imbalances-where cortisol is disproportionately high and DHEA low-have been linked to various health problems.

Subjects will be provided with an at-home saliva collection kit with instructions to collect saliva at four different timepoints throughout the day (waking, Noon, 6pm, before bed), allowing assessment of the body's natural cortisol rhythm (diurnal pattern) and identify potential imbalances related to stress or adrenal gland function.

Stress/Mood/Sleep/Beauty/Focus Assessments Changes in stress/mood/sleep/beauty/focus will be assessed using five research-validated surveys: the Perceived Stress Scale (PSS), Pittsburgh Sleep Quality Index (PSQI), Profile of Mood States (POMS), Beauty Quality of Life survey (BeautyQOL), and the Adult ADHD Self-Report Scale (ASRS). Each survey has been used in numerous clinical trials and their scientific validity is well established (https://psycnet.apa.org/record/2011-08434-004; https://www.tandfonline.com/doi/abs/10.1080/10413200008404210)

The PSS determines how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress, where a higher score indicates a greater level of perceived stress experienced by the individual, with scores typically ranging from 0 (low stress) to 40 (high stress).

The Pittsburgh Sleep Quality Index (PSQI) is a self-reported questionnaire that assesses a person's overall sleep quality over the past month by asking 19 questions categorized into seven components: sleep quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances, sleep medication use, and daytime dysfunction; a higher total score indicates poorer sleep quality, with a score above 5 generally considered indicative of poor sleep (higher scores indicate worse sleep quality).

The POMS questionnaire measures 6 primary psychological factors (tension, depression, anger, fatigue, vigor, or confusion) plus the combined global mood state as an indication of overall subjective well-being. The POMS profile uses 65 adjective-based intensity scales scored on a 0-4 hedonic scale (e.g. "not at all" to "extremely"). The 65 adjective responses are categorized into the 6 mood factors (tension, depression, anger, fatigue, vigor, or confusion), tabulated, scored, and analyzed. The output of the POMS questionnaire is an assessment of the positive and negative moods of each subject at baseline and post-supplementation.

The BeautyQoL instrument, which is composed of 42 questions covering different aspects related to self-perception of beauty, skin health, and Quality of Life and has been validated in 16 languages and 13 countries. The BeautyQoL is specific to physical appearance and is highly sensitive and is capable of capturing even smallest variations in Quality of Life, brought about by the use of innovative cosmetic and beauty care products, or changes in the physical appearance following aesthetic interventions.

The Adult ADHD Self-Report Scale (ASRS) is a tool designed for screening of Attention-Deficit/Hyperactivity Disorder (ADHD) in adults. Developed in collaboration between the World Health Organization (WHO) and researchers at Harvard Medical School, the ASRS consists of 18 items divided into two main domains: inattention and impulsivity.

Product administration instructions:

All subjects will be instructed to follow the same daily protocol to take one capsule (500mg Black Seed Oil or matching Placebo) during a main meal (breakfast, lunch or dinner) with a beverage of their choice. Subjects will be in regular/periodic contact with their coaches and with study monitor, and product compliance will be assessed by measuring unused product at study completion.

Informed Consent An informed consent form (ICF) will be written in accordance with established criteria of the Institutional Review Board (IRB) and the appropriate federal regulations (eg, 21 CFR Parts 50 and 56) to describe the study plan, procedures, and risks. The investigator, the sponsor, and the IRB must all approve the ICF and any ICF amendments or administrative changes before they are used.

Investigators will ensure that each subject is clearly and fully informed of the purpose, potential risks, and requirements of study participation. Written informed consent must be obtained from each subject before performing any screening or other study procedures.

The rights, safety, and well-being of the study subjects are the most important considerations and come before the interests of the study.

Monitoring for Adverse Events An adverse event (AE) is any undesirable symptom or occurrence experienced by a subject during a clinical trial. It may or may not be considered related to the study product. Assessment of an adverse event (AE) involves: subjective reports from the subject, observation by members of the research team and clinically significant abnormal laboratory results.

AE severity (intensity) will be classified as mild, moderate, or severe according to the following definitions:

* Mild: causing no limitation in normal activities
* Moderate: causing some limitation in normal activities
* Severe: causing significant limitation in or the inability to perform normal activities.

The PI will assess and assign the severity of all reported AE's.

The PI is responsible for determining the relationship between an AE and the study products. The relationship will be classified as one of the following:

* Probable: good reasons and sufficient documentation to assume a causal relationship
* Possible: a causal relationship is conceivable and cannot be dismissed
* Unlikely: the event is most likely related to an etiology other than the trial product
* Definitely not related: the event is not related to the study product

All SAE's will also be reported to the IRB within 24 hours of site knowledge using IRB requirements and guidelines. It is the sponsor's decision whether or not an SAE should be reported to the Food and Drug Administration (FDA).

Data Management & Analysis Data will be recorded onto case report forms (CRFs) by 3 Waves Wellness staff and will be entered into Excel worksheets. The computerized data will be anonymized; subject identifiers will be limited to ID numbers and subject initials. Data files will be retained in a physically secure location, and regular backup copies will be created and stored in a separate secure location. Prior to analysis, 3 Waves Wellness staff will review all data, comparing the values in the data files with the values on the original CRFs, and correcting any discrepancies found.

All data elements will be evaluated for reasonableness and consistency, and any suspicious or impossible values will be referred back to source documents for verification or correction.

The final data will be analyzed separately (each subject cohort compared to placebo) and combined (both subject cohorts compared to placebo). Data will be analyzed by the Per-Protocol (PP) method - consisting of all subjects who completed all scheduled visits, had no protocol deviations that (in the judgment of the principal investigator) would have invalidated their efficacy data, and were between 80 and 120% compliant with the specified product dosing. If a subject is only slightly outside the allowable compliance limits, the principal investigator can include that subject in the PP population. If the overall compliance is not available for one of the testing phases of the study (e.g. if the subject has forgotten to return the unused product), the PI can make a determination of compliance based on the 3 Waves Wellness staff's familiarity with the subject or on the subject's compliance during the other testing phase(s) of the study.

The efficacy endpoints will be tested using an analysis of variance (ANOVA) and pairwise test between the product group (active product or placebo) and variable of interest (Cortisol, POMS, etc). As this is not a Phase III FDA drug study, each comparison will be considered an independent question of interest, and each comparison will be interpreted at the test-wise 0.05 alpha level (p≤0.05 will be considered significant).

ELIGIBILITY:
Inclusion Criteria:

* • Healthy moderately-stressed adults; Female and Male / Age 18-70

  * Informed consent
  * Ability/desire to participate in 8-week supplement program

Exclusion Criteria:

* Inability to complete prescribed supplement regimen
* Current use of incompatible medications or supplements, including anti-inflammatory or antidepressant medications and supplements in the last 4 weeks before the study and during the study
* Auto-immune or inflammatory disease diagnosis
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
cortisol | from baseline until week 8, with interim measures at week 1 and week 4
  measures of salivary cortisol

SECONDARY OUTCOMES:
mood state | from baseline to week 8, with interim measures at week 1 and week 4
  Subjective assessments of psychological mood state using five research-validated surveys: the Perceived Stress Scale (PSS), Pittsburgh Sleep Quality Index (PSQI), Profile of Mood States (POMS), Beauty Quality of Life survey (BeautyQOL), and the Adult ADHD Self-Report Scale (ASRS). Each survey has been used in numerous clinical trials and their scientific validity is well established.

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Talbott, PhD, Principal Investigator — 3 Waves Wellness
Locations (1):
- 3 Waves Wellness, Plymouth, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No